CLINICAL TRIAL: NCT04526951
Title: TENecteplase in Central Retinal Artery Occlusion Study (TenCRAOS): A Randomized Placebo-controlled Trial of Early Systemic Tenecteplase Treatment in Patients With Central Retinal Artery Occlusion.
Brief Title: TENecteplase in Central Retinal Artery Occlusion Stuy (TenCRAOS)
Acronym: TenCRAOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anne Hege Aamodt, Professor, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Oslo UH; 2018-002546-36 (EudraCT Number); 2019/327 (Other: Ethics Committee in Norway); 2024-517606-29-00 (EU CTIS Number)
Record Dates: First submitted 2020-08-20; First posted 2020-08-26 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-06

CONDITIONS: Central Retinal Artery Occlusion
Keywords: thrombolysis tenecteplase
MeSH Terms: conditions — Retinal Artery Occlusion | interventions — Tenecteplase; Aspirin

STUDY DESIGN:
Intervention Model Description: A prospective, randomized-controlled, double-dummy, double-blind phase 3 multi-centre trial of TNK 0.25 mg/kg + placebo vs. ASA + placebo (2 arms with 1:1 block randomisation). At all participating centers, ophthalmologists are involved in the diagnosis and visual outcome measurements using a standardized protocol. The patients will be promptly examined by the ophthalmologist. As soon as the CRAO is diagnosed by the ophthalmologist, the patients will be managed in the stroke unit during treatment, monitoring, and medical investigations. After treatment in the stroke unit, the patients will be re-examined by an ophthalmologist and a neurologist as an out-patient at (30 ±5) and 90 (±15) days.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tenecteplase (Active Comparator): The total dose of tenecteplase is 0.25 mg/kg body weight, maximum 25 mg. The total dose will be given as an intravenous bolus
  Interventions: Drug: Intravenous injection of Tenecteplase and one dose of placebo tablet
- acetylsalicylic acid (Active Comparator): one tablet of aspirin 300 mg Other Name: Aspirin
  Interventions: Drug: One tablet of Acetylsalicylic Acid and one dose of IV placebo

INTERVENTIONS:
Drug: Intravenous injection of Tenecteplase and one dose of placebo tablet — Drug: Tenecteplase Tenecteplase administered as an intravenous injection (0.25 mg/kg body weigh; maximum 25 mg)
  Other Names: Metalyse
  Arms: Tenecteplase
Drug: One tablet of Acetylsalicylic Acid and one dose of IV placebo — 300 mg Acetylsalisylic acid
  Other Names: Aspirin
  Arms: acetylsalicylic acid

SUMMARY:
TENecteplase in Central Retinal Artery Occlusion (TenCRAOS): A Prospective, randomized-controlled, double-dummy, double-blind phase 3 multi-centre trial of TNK 0.25 mg/kg + placebo vs. ASA + placebo (2 arms with 1:1 block randomization).

A Prospective, randomized-controlled, double-dummy, double-blind phase 3 multi-centre trial of TNK 0.25 mg/kg + placebo vs. ASA + placebo (2 arms with 1:1 block randomization). At all participating centers, ophthalmologists are involved in the diagnosis and visual outcome measurements using a standardized protocol. The patients will be promptly examined by the ophthalmologist. As soon as the CRAO is diagnosed by the ophthalmologist, the patients will be managed in the stroke unit during treatment, monitoring, and medical investigations. After treatment in the stroke unit, the patients will be re-examined by an ophthalmologist and a neurologist as an out-patient at (30 ±5) and 90 (±15) days

DETAILED DESCRIPTION:
Central retinal artery occlusion (CRAO) is an ophthalmologic emergency that, without prompt revascularization, bears high risk of permanent blindness. The condition is typically the result of an artery-to-artery embolism from a carotid plaque or cardio embolism. A recent meta-analysis of observational data indicates that prompt revascularization with systemic thrombolysis might improve outcome. A randomized controlled trial of early systemic thrombolysis for CRAO is therefore warranted. The aim of this project is to assess the effect of systemic tissue plasminogen activator tenecteplase versus placebo administered within 4.5 hours of CRAO onset in patients admitted to the participating hospitals in Europe. The main endpoint is the proportion of patients with ≤ 0.7 logMAR visual acuity 30 (±5) days after treatment, representing an improvement in visual acuity of at least 0.3 logMAR, equal to at least 15 letters/three lines on a visual acuity chart. In addition, we will access differences in visual field parameters and patient reported outcome measures between the groups. This study is based on a broad collaboration and interaction between leading ophthalmologists and neurologists in European centres.

ELIGIBILITY:
Inclusion Criteria:

1. Non-arteritic central retinal artery occlusion with ≥ 1.0 logMAR visual acuitiy and symptoms lasting less than 4.5 hours.
2. Ability to administer the Investigator Medicinal Product (IMP) within 4.5 hours of symptom onset.
3. Age ≥18 years.
4. Informed written consent of the patient.
5. A woman of childbearing potential (WOCBP) must confirm that in her opinion, she cannot be pregnant, OR if there is a possibility that she is pregnant, a negative pregnancy test must be confirmed before any IMP is given.

Exclusion Criteria:

1. Other active intervention targeting CRAO.
2. Branch retinal artery occlusion, cilioretinal artery supplying the macula, combined arterial-venous occlusion, proliferative diabetic retinopathy, elevated intraocular pressure (> 30 mmHg) or clinical suspicion of ophthalmic artery occlusion occlusion (e.g. choroidal nonperfusion, absence of cherry red spot, no light perception).
3. Systemic diseases; severe general diseases, systemic arterial hypertension (blood pressure >185/110 mmHg), despite medical therapy, or clinical suspicion of acute systemic inflammation.
4. Presence of intracranial haemorrhage on brain MRI/CT.
5. Medical history: heart attack within the last 6 weeks, intracerebral bleeding or neurosurgical operation within the last 4 weeks, therapy with anticoagulation, allergic reaction to contrast agent, hemorrhagic diathesis, aneurysms, inflammatory vascular diseases (eg, giant cell arteritis, granulomatosis with polyangitis), endocarditis, or gastric ulcer.
6. No willingness and ability of the patient to participate in all follow-up examinations.
7. Pregnancy (if suspicion of pregnancy s-hCG or u-hCG must be negative).
8. Allergy or intolerance to any ingredients of IMP or placebo or gentamicin.
9. Other conditions / circumstances likely to lead to poor treatment adherence (eg, history of poor compliance, alcohol or drug dependency, no fixed abode).
10. Significant bleeding disorder either at present or within the past 6 months.
11. Effective oral anticoagulant treatment, eg, warfarin sodium (INR >1.3).
12. Effective anticoagulant treatment with heparin or low molecular weight heparin the last 48 hours.
13. Any history of central nervous system damage (ie, neoplasm, aneurysm, intracranial or spinal surgery).
14. Known hemorrhagic diathesis.
15. Major surgery, biopsy of a parenchymal organ, or significant trauma within the past 2 months (this includes any trauma associated with acute myocardial infarction).
16. Recent non-compressible vessel puncture within 2 weeks.
17. Recent trauma to the head or cranium.
18. Prolonged cardiopulmonary resuscitation (>2 minutes) within the past 2 weeks.
19. Acute pericarditis and/or subacute bacterial endocarditis.
20. Acute pancreatitis.
21. Severe hepatic dysfunction, including hepatic failure, cirrhosis, portal hypertension (oesophageal varices) and active hepatitis.
22. Active peptic ulceration.
23. Arterial aneurysm and known arterial/venous malformation.
24. Neoplasm with increased bleeding risk.
25. Any known history of hemorrhagic stroke or stroke of unknown origin.
26. Known history of ischemic stroke or transient ischemic attack in the preceding 3 months.
27. Dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with ≤ 0.7 logMAR visual acuity in the affected eye at 30 (±5) days after treatment, representing an improvement in visual acuity of at least 0.3 logMAR (intention-to-treat (ITT) analysis). | 30 (±5) days
  logMAR

SECONDARY OUTCOMES:
Proportion of patients with ≤ 0.5 logMAR visual acuity in the affected eye at 30 (±5) and 90 (±15) days. | 30 (±5) and 90 (±15) days
  logMAR
Mean improvement in logMAR visual acuity in the affected eye from baseline to 30 (±5) and 90 (±15) days. | 30 (±5) and 90 (±15) days
  logMAR
Proportion of patients with visual recovery (logMAR ≤ 0.7) and (logMAR ≤ 0.5) in the affected eye 30 (±5) and 90 (±15) days in patients who were treated with tenecteplase within 3 hours of onset | 30 (±5) and 90 (±15) days
  logMAR
Number of test points seen (of 100) on monocular Esterman perimetry at 30 (±5) and 90 (±15) days | 30 (±5) and 90 (±15) days
  Number of test points
Acute ischemic lesions on follow-up on diffusion-weighted (DWI) MRI or on brain CT at baseline and 24hrs. | 24 hours
  DWI lesions
National Institutes of Health Stroke Scale score (NIHSS) at 24hrs and discharge. | 24 hours
  NIHSS score
Modified Rankin Scale score (mRS) at discharge, 30 (±5) and 90 days (±15) days. | Discharge, 30 (±5) and 90 days (±15) days.
  mRS score
Mean score on National Eye Institute Visual Function Questionnaire (NEI-VFQ 25) at 30 (±5) and 90 (±15) days | 30 (±5) and 90 (±15) days
  Visual function related quality of life at 30 and 90 days. Measures the dimensions of self-reported vision-targeted health status that are most important for persons who have chronic eye diseases. 100 = best possible, 0 = worst possible
Mean score on EQ-5D at 30 (±5) and 90 (±15) days | 30 (±5) and 90 (±15) days
  Quality of life reported at 30 and 90 days. Health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Presence of ocular neovascularisation at 30 (±5) and 90 (±15) days | 30 (±5) and 90 (±15) days
  presence

OTHER OUTCOMES:
All-cause and stroke-related death at discharge, 30 (±5) and 90 (±15) days. | Discharge assessed up to 7 days , 30 (±5) and 90 (±15) days
  Mortality
Proportion of patients with any intracranial haemorrhage at 24 hrs | 24 hours
  Intracranial haemorrhage
Proportion of patients with symptomatic intracranial haemorrhage until discharge. | at discharge, assessed up to 7 days
  Symptomatic intracranial haemorrhage
Proportion of patients with complications such as systemic bleeding at 24 hrs, discharge and 30 (±5) days | 24 hours, at discharge assessed up to 7 days and 30 (±5) days
  Systemic bleeding
Other serious adverse events | 24 hours, at discharge, 30 (±5) days and 90 days (±15) days.
  Frequency of serious adverse events
Occurrence of adverse events | 24 hours, at discharge assessed up to 7 days, 30 (±5) days and 90 days (±15) days.
  Frequency of adverse events
Retrobulbar spot sign detection using Duplex/Doppler ultrasound at baseline, point-of-care ultrasound (POCUS) | 30 (±5) and 90 (±15) days
  Frequency of retrobulbar spot sign
Retrobulbar spot sign and central retinal artery recanalisation using Duplex/Doppler ultrasound at 24h and discharge | 24 hours and at discharge assessed up to 7 days
  Frequency of retrobulbar spot sign
Macular optical coherence tomography (OCT) volume scans and macular OCT angiography (OCT-A) at 30 and 90 days | 30 (±5) and 90 (±15) days
  OCT measures

CONTACTS AND LOCATIONS:
Locations (18):
- Belgium (2):
  - University Hospital Antwerp, Antwerp
  - University Hospital Leuven, Leuven
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Bispebjerg University Hospital, Copenhagen
  - Rigshospitalet University Hospital, Copenhagen
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Turku University Hospital, Turku
- Lithuania (2):
  - Kauno Klinikos Kaunas, Kaunas
  - Vilnius University Hospital, Vilnius
- Norway (8):
  - Haukeland University Hospital, Bergen
  - Vestre Viken Hospital Trust Drammen, Drammen
  - Østfold Hospital Trust Kalnes, Dept of Ophthalmology, Grålum
  - Helse Nord Trøndelag Trust, Namsos
  - Oslo University Hospital, Oslo
  - Telemark Hospital Trust, Skien
  - St Olav University Hospital, Trondheim
  - Vestfold Hospital Trust, Tønsberg
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to share data with the THEIA trial and REVISION trial for IPD meta analysis
Supporting Information: Study Protocol, ICF
Time Frame: Protocol is planned to be published in peer-reviewed journal in 2023
Access Criteria: Protocol is planned to be published in peer-reviewed journal in 2023 and will be available at the journal site

REFERENCES:
- [Derived] Ryan SJ, Jorstad OK, Skjelland M, Pesonen M, Simonsen CZ, Bek T, Blauenfeldt RA, Ijas P, Laitinen A, Khanevski A, Krohn J, Rodahl E, Lemmens R, Demeestere J, Cassiman C, Nakstad I, Evensen K, Sandell T, Hamann S, Truelsen TC, Christensen LM, Rosenbaum S, Matijosaitis V, Zemaitiene R, Ellekjaer H, Almaas E, Austeng D, Mazya MV, Traisk F, Ylikotila P, Salmi U, Jenssen KN, Lisether H, Breivik C, Devik K, Honningsvag LE, Valaikiene J, Cimbalas A, Malmberg VN, Anderson E, Roy A, Skattor TH, Kraglund KL, Kefaloykos C, Olsen IC, Vanacker P, Strbian D, Moe MC, Aamodt AH; TenCRAOS Investigators. A Randomized Trial of Tenecteplase in Acute Central Retinal Artery Occlusion. N Engl J Med. 2026 Jan 29;394(5):442-450. doi: 10.1056/NEJMoa2508515. PMID 41604638